CLINICAL TRIAL: NCT00893932
Title: Leptin: a Therapeutic Option for Treating Catabolic States and Malnutrition in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sigal Sviri MD, Hadassah Medical Organization
Other Study IDs: LeptinHadassahMO
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-04

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: SIRS leptin outcome sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for leptin levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SIRS

SUMMARY:
Leptin is a hormone that plays a central role in food intake and energy balance. It is secreted by fat cells, released into the circulation and transported into the central nervous system (brain), where it regulates energy balance and food intake. The overall effects of leptin appear to reduce food intake when the body is calorically satisfied, and to alter metabolic rate A decrease in the amount of body fat, which occurs after fasting, reduces the level of leptin, thereby stimulating food intake. Systemic Inflammation is a condition in which body tissues respond to stress. It may be associated with severe infection or other stimuli such as trauma, and may lead to organ failure and death. It has been shown, that Leptin may be a "survival protein", where higher levels are associated with lower mortality. The investigators set out to quantify the levels of Leptin in critically ill patients in association with other markers of inflammation and mortality.

DETAILED DESCRIPTION:
Patients admitted to the Medical Intensive Care Unit who comply with criteria for SIRS (Systemic inflammatory response syndrome) will be enrolled into the study.

SIRS can be diagnosed when two or more of the following are present:

* Heart rate > 90 beats per minute
* Body temperature < 36 or > 38°C
* Hyperventilation (high respiratory rate) > 20 breaths per minute or, on blood gas, a PaCO2 < 32 mm Hg or mechanically ventilated
* White blood cell count < 4000 cells/mm3 or > 12000 cells/mm3 (< 4 x 109 or > 12 x 109 cells/L), or the presence of greater than 10% immature neutrophils.

Clinical parameters will be collected including: demographics, diagnosis, past medical history, past and present medications, fluids and nutrition administered, oxygenation and ventilation parameters, hemodynamic status and renal function and/or replacement therapy. Severity of illness using APACHE II score, major events during unit stay such as procedures, length of inotropic support, complications. Length of unit and hospital stay, length of ventilation, unit and hospital outcome.

Baseline leptin levels (within 8 hours of admission) will be obtained. Subsequent levels of leptin will be measured every 2 days or until discharge from the unit or death.

Serial blood count, chemistry, total protein, albumin, renal and liver function, glucose and insulin levels, lactate, total cholesterol, TSH, T3, IL-6, TNF-a, adiponectin, CRP, ESR, urine output, creatinine clearance and Nitrogen balance will be obtained.

ELIGIBILITY:
Inclusion Criteria:All patients with Systemic Inflammatory Response Syndrome (SIRS).

SIRS can be diagnosed when two or more of the following are present:

* Heart rate > 90 beats per minute
* Body temperature < 36 or > 38°C
* Hyperventilation (high respiratory rate) > 20 breaths per minute or, on blood gas, a PaCO2 < 32 mm Hg or mechanically ventilated
* White blood cell count < 4000 cells/mm3 or > 12000 cells/mm3 (< 4 x 109 or > 12 x 109 cells/L), or the presence of greater than 10% immature neutrophils.

Exclusion Criteria:

* Patients under 18, pregnant patients, patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Medical ICU and diagnosed with SIRS
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To assess in the intensive care setting leptin levels and their relationship to inflammatory cytokines during the course of catabolic illnesses and following recovery. | 14 days, discharge from ICU or death

SECONDARY OUTCOMES:
To measure indices of metabolism, catabolism and ICU outcome and their associations with leptin response. | 14 days, ICU discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Sviri, MD, Principal Investigator — Hadassah Medical Organization; Yosepha Avraham, pHD, Principal Investigator — Hebrew University
Locations (1):
- Medical ICU, Hadassah Medical Organization, Jerusalem, Israel